CLINICAL TRIAL: NCT02267382
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging Study to Evaluate the Efficacy and Safety of VT-1161 Oral Tablets in the Treatment of Patients With Recurrent Vulvovaginal Candidiasis
Brief Title: A Study to Evaluate Oral VT-1161 in the Treatment of Patients With Recurrent Vaginal Candidiasis (Yeast Infection)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Viamet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: VMT-VT-1161-CL-006
Record Dates: First submitted 2014-10-08; First posted 2014-10-17 (Estimated); Results first posted 2019-10-04 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Recurrent Vulvovaginal Candidiasis
MeSH Terms: conditions — Candidiasis, Vulvovaginal | interventions — VT-1161

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- VT-1161 Low-dose 3-month (Experimental): 1 VT-1161 150mg tablet and 1 placebo tablet once daily for 7 days, then once weekly for 11 weeks, followed by 2 placebo tablet once weekly for 12 weeks
  Interventions: Drug: VT-1161
- VT-1161 Low-dose 6-month (Experimental): 1 VT-1161 150mg tablet and 1 placebo tablet once daily for 7 days, then once weekly for 23 weeks
  Interventions: Drug: VT-1161
- VT-1161 High-dose 3-month (Experimental): 2 VT-1161 150mg tablets once daily for 7 days, then once weekly for 11 weeks, followed by 2 placebo tablet once weekly for 12 weeks
  Interventions: Drug: VT-1161
- VT-1161 High-dose 24-week (Experimental): 2 VT-1161 150mg tablets once daily for 7 days, then once weekly for 23 weeks
  Interventions: Drug: VT-1161
- Placebo (Placebo Comparator): 2 placebo tablets once daily for 7 days, then once weekly for 23 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VT-1161
  Arms: VT-1161 High-dose 24-week; VT-1161 High-dose 3-month; VT-1161 Low-dose 3-month; VT-1161 Low-dose 6-month
Drug: Placebo
  Arms: Placebo

SUMMARY:
VT-1161 is a novel, oral inhibitor of fungal lanosterol demethylase (CYP51). In vitro and in vivo pharmacology studies have demonstrated that VT-1161 is highly active against Candida albicans and also non-albicans Candida species that cause vulvovaginal candidiasis. VT-1161 is highly selective for fungal CYP51, and data suggests that it may avoid the side-effect profile that limits the use of commonly prescribed antifungal agents for the treatment of recurrent yeast infections.

ELIGIBILITY:
Key Inclusion Criteria:

Clinical diagnosis of symptomatic acute VVC

3 or more episodes of acute VVC in the past 12 months

Positive KOH

Minimum composite vulvovaginal signs and symptoms score of ≥3 at Screening

Composite vulvovaginal signs and symptoms score of <3 at Baseline

Must be able to swallow tablets

Key Exclusion Criteria:

Evidence of major organ system disease

Presence or a history of another vaginal or vulvar condition(s)

History of cervical cancer

Poorly controlled diabetes mellitus

Pregnant

Recent use of topical or systemic antifungal drugs

Recent use of immunosuppressive or system corticosteroid therapies

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2015-02-10 (Actual); Primary Completion 2016-11-09 (Actual); Study Completion 2016-11-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (31):
- United States (31):
  - University of Alabama Birmingham, Birmingham, Alabama
  - Precision Trials, Phoenix, Arizona
  - NEA Baptist Clinic, Jonesboro, Arkansas
  - Axis Clinical Trials, Los Angeles, California
  - Genesis Center for Clinical Research, San Diego, California
  - Altus Research, Lake Worth, Florida
  - Healthcare Clinical Data, Miami, Florida
  - Community Medical Research, North Miami, Florida
  - Vision Clinical Research, Palm Beach, Florida
  - Physician Care Clinical Research LLC, Sarasota, Florida
  - Clinical Research of West Florida, Tampa, Florida
  - Cypress Medical Research Center, Wichita, Kansas
  - Clinical Trials Management LLC, Covington, Louisiana
  - Clinical Trials Management LLC, Metairie, Louisiana
  - New England Center for Clinical Research, Fall River, Massachusetts
  - Clinical Research of Nevada, Las Vegas, Nevada
  - R. Garn Mabey, Jr. M.D. Chartered, Las Vegas, Nevada
  - OB/GYN Clinical Research, Lawrenceville, New Jersey
  - Women's Health Research Center, Plainsboro, New Jersey
  - Suffolk OB-GYN, Port Jefferson, New York
  - United Women's Clinical Research-Raleigh, Raleigh, North Carolina
  - Lyndhurst Clinical Research, Winston-Salem, North Carolina
  - Radiant Research, Akron, Ohio
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - Magee Women's Hospital, Pittsburgh, Pennsylvania
  - Brownstone Clinical Trials, Fort Worth, Texas
  - TMC Life Research, Houston, Texas
  - Brownstone Clinical Trials, Irving, Texas
  - Clinical Trials of Texas, San Antonio, Texas
  - Physician's Research Options LLC, Sandy City, Utah
  - Seattle Women's Health Research Gynecology, Seattle, Washington

REFERENCES:
- [Derived] Vanreppelen G, Nysten J, Baldewijns S, Sillen M, Donders G, Van Dijck P. Oteseconazole (VIVOJA) for prevention of recurrent vulvovaginal candidiasis. Trends Pharmacol Sci. 2023 Jan;44(1):64-65. doi: 10.1016/j.tips.2022.10.004. Epub 2022 Nov 14. No abstract available. PMID 36396498
- [Derived] Brand SR, Degenhardt TP, Person K, Sobel JD, Nyirjesy P, Schotzinger RJ, Tavakkol A. A phase 2, randomized, double-blind, placebo-controlled, dose-ranging study to evaluate the efficacy and safety of orally administered VT-1161 in the treatment of recurrent vulvovaginal candidiasis. Am J Obstet Gynecol. 2018 Jun;218(6):624.e1-624.e9. doi: 10.1016/j.ajog.2018.03.001. Epub 2018 Mar 11. PMID 29534874

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 254 subjects were enrolled in the 14-day open-label Induction Phase of the study after providing consent. Those subjects whose acute VVC infections resolved during the Induction Phase (a total of 215) entered the Maintenance Phase of the study.
Period: Overall Study
Arm/Group | VT-1161 Low-dose 3-month | VT-1161 Low-dose 6-month | VT-1161 High-dose 3-month | VT-1161 High-dose 24-week | Placebo
Started | 42 | 43 | 43 | 41 | 46
Completed | 35 | 33 | 34 | 35 | 39
Not Completed | 7 | 10 | 9 | 6 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VT-1161 Low-dose 3-month | VT-1161 Low-dose 6-month | VT-1161 High-dose 3-month | VT-1161 High-dose 24-week | Placebo | Total
Number analyzed (Participants) | 42 | 43 | 43 | 41 | 46 | 215
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.0 (10.2) | 34.6 (9.09) | 34.2 (9.28) | 33.8 (10.13) | 35.4 (11.2) | 34.6 (9.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 43 | 43 | 41 | 46 | 215
  Male | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Subjects With 1 or More Culture-verified Acute VVC Episodes Through Week 48 of the Study in the Intent-to-treat Population.
Description: A culture-verified acute VVC episode was defined as a positive fungal culture for Candida species associated with a clinical signs and symptoms score of ≥3. To calculate the 'signs and symptoms' score, each vulvovaginal sign (erythema, edema, excoriation) and symptom (itching, burning, irritation) was scored using the following scale, with higher scores indicating a worse outcome.
  0 = none (complete absence of any sign or symptom)
  1. = mild (slight)
  2. = moderate (definitely present)
  3. = severe (marked, intense)
Time Frame: 48 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | VT-1161 Low-dose 3-month | VT-1161 Low-dose 6-month | VT-1161 High-dose 3-month | VT-1161 High-dose 24-week | Placebo
Number analyzed (Participants) | 42 | 43 | 43 | 41 | 46
Participants | 2 | 3 | 0 | 2 | 24

ADVERSE EVENTS:
Description: Safety analyses were performed on the subjects in the safety population, which was defined as all subjects who were randomly assigned to VT-1161 or placebo and received at least 1 dose of study drug. Subjects were analyzed according to the treatment regimen received, regardless of the treatment regimen to which they were randomly assigned.
Arm/Group | VT-1161 Low-dose 3-month | VT-1161 Low-dose 6-month | VT-1161 High-dose 3-month | VT-1161 High-dose 24-week | Placebo
Serious Adverse Events (participants affected / at risk) | 1/41 | 0/42 | 1/42 | 2/41 | 1/45
Other Adverse Events (participants affected / at risk) | 26/41 | 31/42 | 30/42 | 28/41 | 35/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VT-1161 Low-dose 3-month (N=41) | VT-1161 Low-dose 6-month (N=42) | VT-1161 High-dose 3-month (N=42) | VT-1161 High-dose 24-week (N=41) | Placebo (N=45)
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Meningitis viral (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VT-1161 Low-dose 3-month (N=41) | VT-1161 Low-dose 6-month (N=42) | VT-1161 High-dose 3-month (N=42) | VT-1161 High-dose 24-week (N=41) | Placebo (N=45)
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 3 | 2 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Abdominal tenderness (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 1
Dental carries (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 2 | 1 | 1 | 1
Esophageal stenosis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Esophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 3 | 2 | 2 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 0
Device breakage (General disorders) | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 2 | 1 | 0 | 1
Influenza-like illness (General disorders) | 0 | 1 | 0 | 0 | 0
Mass (General disorders) | 0 | 0 | 1 | 0 | 0
Pain (General disorders) | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0
Ulcer (General disorders) | 0 | 0 | 1 | 0 | 0
Food allergy (Immune system disorders) | 0 | 0 | 0 | 1 | 0
Rubber sensitivity (Immune system disorders) | 0 | 1 | 0 | 0 | 0
Acute sinusitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Bacterial infection (Infections and infestations) | 0 | 2 | 1 | 0 | 1
Bacterial vaginosis (Infections and infestations) | 7 | 6 | 7 | 1 | 9
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Bronchopneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Chlamydial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Ear infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Escherichia vaginitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Eye infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Fungal skin infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 2 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Genital herpes (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Helicobacter infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Hordeolum (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 3 | 1 | 0
Laryngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Meningitis viral (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 2 | 4 | 3 | 0
Oropharyngeal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Papilloma viral infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Perineal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Perirectal abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 5 | 6 | 3 | 2 | 3
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Streptococcal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 2
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Tinea infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Tooth infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Trichomoniasis (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 3 | 2 | 1 | 2
Urinary tract infection (Infections and infestations) | 4 | 4 | 6 | 7 | 10
Vaginitis bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Vulvitis (Infections and infestations) | 0 | 1 | 0 | 1 | 1
Wound infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 2 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Mountain sickness acute (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 3 | 0 | 0 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Vaginal laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 1 | 0 | 0
Smear cervix abnormal (Investigations) | 1 | 0 | 0 | 0 | 0
Ureaplasma test positive (Investigations) | 1 | 0 | 0 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 2 | 2 | 0
Fibroadenoma of breast (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
7th nerve paralysis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Cervical radiculopathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 1 | 0
Headache (Nervous system disorders) | 5 | 0 | 2 | 2 | 5
Hypoesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Tension headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0
Vomiting in pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 1 | 1 | 0
Depressed mood (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0
Cystitis interstitial (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 1 | 2 | 0
Micturition urgency (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Stress urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Urine odor abnormal (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Adnexa uteri pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Amenorrhea (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 1
Breast mass (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 1
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 1
Breast tenderness (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Cervix disorder (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Dysmenorrhea (Reproductive system and breast disorders) | 1 | 0 | 0 | 1 | 0
Dyspareunia (Reproductive system and breast disorders) | 1 | 0 | 0 | 1 | 0
Edema genital (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Menopausal symptoms (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 1
Menstrual disorder (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 2 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 2
Polycystic ovaries (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Postmenopausal hemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Uterine enlargement (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Uterine tenderness (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Vaginal discharge (Reproductive system and breast disorders) | 1 | 0 | 0 | 1 | 1
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 | 1 | 1 | 0 | 0
Vaginal odor (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Vulvovaginal burning sensation (Reproductive system and breast disorders) | 1 | 1 | 1 | 0 | 1
Vulvovaginal discomfort (Reproductive system and breast disorders) | 3 | 2 | 0 | 0 | 2
Vulvovaginal disorder (Reproductive system and breast disorders) | 1 | 0 | 1 | 0 | 0
Vulvovaginal dryness (Reproductive system and breast disorders) | 2 | 0 | 1 | 0 | 0
Vulvovaginal erythema (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 2 | 1 | 2 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0
Miliaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Neurodermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Pruritis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 3 | 0 | 1
Seborrheic dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 2 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Neither Institution nor Principal Investigator shall publish the results of the Trial without the prior written consent of Sponsor, which it may withhold in its sole discretion.